CLINICAL TRIAL: NCT07248449
Title: Effects of Cuevas Medak Exercises Vs Rebound Exercises on Physical Fitness in Children With Down Syndrome
Brief Title: Physical Fitness in DS: A Comparison of Cuevas Medak and Rebound Exercises
Acronym: DownSyndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/AYESHAAFZAL
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Down Syndrome
Keywords: Cuevas Medek Exercise, Rebound Exercise, Down syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial (RCT) designed to compare the effectiveness of two different exercises, Cuevas Medak Vs Rebound Exercises on physical Fitness of Down Syndrome. The study will involve 22 participants of both gender between the ages of 3-8 years. These participants will be randomly divided into two groups. children who will be able to understand the commands given to them. Using lottery method, the participants will be randomly divided into two groups. One group will be given Cuevas Medek Exercises and the other with Rebound exercises. SAMU-Disability Fitness (DISFIT) battery will be used to assess the Physical Fitness in Down syndrome. Both groups will be given three treatment session per week for 12 weeks and total time for each session will be 30-45 minutes. Data will be analyzed by using SPSS v 26.Sample size is 22 and is calculated by epitol
Who Masked: Participant
Masking Description: Participants will get separate treatment protocol and possible efforts will be put to mask the both groups about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental:11 children of DS will be given Cuevas Medak Exercises for 12 weeks (Experimental): Baseline treatment will be applied to patient through following functional activities. Core strengthening exercises (isometrics) shall be given as a common treatment. This involved completing two sets of 15 repetitions with each repetition held for 5 seconds. The children in group 1 received Cuevas Medek exercise 3 times per week for 3 successive months. The patient was supported at board at the leg level with slight posterior support to maintain balance. After being lifted off the ground for a few seconds, gentle up and down oscillations were applied. The study utilized three wooden boxes with identical dimensions measuring 20cm x 40cm x 60cm each, along with a larger box, a wooden plate, and two planks of equal size measuring 17cm x 80cm. These items were arranged in various configurations to create structures such as slides, piano flaps, and stairs.
  Interventions: Other: Cuevas Medak Exercises
- Expermental:11 children of DS will be given Rebound Exercises for 15 min (Experimental): Group b will receive Rebound exercise. Baseline treatment will be applied to patient. The children in group 2 received rebounding exercise 3 times per week for 3 successive months. Mini trampoline.Each rebounding session consisted of the following schedule: (3 min of rebounding) - (3 min rest) - (3 min of rebounding) - (3 min rest) - (3 min of rebounding). Thus, one treatment session corresponded to 9 min of rebounding exercise (21). side sitting and high kneeling); bouncing and / or being bounced without leaving the surface of the trampoline.
  Interventions: Other: Cuevas Medak Exercises

INTERVENTIONS:
Other: Cuevas Medak Exercises — Group A 11 children of DS will be given Cuevas Medak Exercises for 12 weeks and total time for each session will be 30-45 min. Group B 11 children of DS will be given Rebound Exercises for 15 min though this can be broken into multiple 3-5 min
  Other Names: Rebound Exercises

SUMMARY:
This randomized clinical trial investigates the comparative effects of Cuevas Medak Exercises Vs Rebound Exercises on physical fitness in DS. The.current study will be single blinded randomized clinical design in which nonprobability convenience sampling technique will be used. Inclusion criteria will be Down Syndrome. both genders will be included. The study involves 22 DS aged 3-8, will be assigned using lottery method, the participants will be randomly divided into two groups. One group will be given Cuevas Medek Exercises and the other with Rebound exercises. SAMU-Disability Fitness (DISFIT) battery will be used to assess the Physical Fitness in Down syndrome. Both groups will be given three treatment session per week for 12 weeks and total time for each session will be 30-45 minutes.

. Data will be analyzed through SPSS version 26.0

DETAILED DESCRIPTION:
Down syndrome is usually associated with developmental delays, mild to moderate intellectual disability, and characteristic physical features. Children with DS usually encounter problems with the motor function as a result of decreased muscle tone, ligamentous laxity, decreased muscle strength, and endurance.

Children with DS experience decreased balance capacity on account of the brain stem and cerebellar hypoplasia leading to disruption of motor function and postural control. DS children have difficulty preserving their body posture which is frequently combined with an abnormality in gait pattern Cuevas Medek Exercises (CME) is a psychomotor therapy approach for rehabilitation programs that involves automatic motor reactions using exercises against gravity provoking the postural control and also describe its neuroplastic outcome. MEDEK is an acronym for a Spanish phrase means "Dynamic Method for Kinesthetic Stimulation infuriating postural control, which is not self-produced due to impaired central nervous system. The main mechanism is to generate new neuronal networks in affected central nervous system by utilizing scientific parameters associated to neuroplasticity (such as repetition, ROM, weight bearing, progression, significant exercises). Down syndrome might be particularly susceptible to loss of basic function because of poor physical fitness. Rebounding exercises are a series of movements based on trampoline exercises, have been used for children with different physical and intellectual disabilities. The Health Bounce, this is a basic movement that involves bouncing up and down on the trampoline.

Rebounding from quality mini trampoline provides all the benefits of other aerobic exercise without the stress impact .The objective of current study is to check the effects of Cuevas Medek exercise VS rebound exercise on physical fitness in children with Down syndrome . The current study will be single blinded randomized clinical design in which nonprobability convenience sampling technique will be used. Inclusion criteria will be Down Syndrome Age ranges between 3-8 yrs, both genders will be included, children who will be able to understand the commands given to them.

Exclusion Criteria will be Patients with medical condition, contracture, musculoskeletal disorders, Atlanta 3 CUEVAS MEDEK EXERCISES VS REBOUND EXERCISES IN DOWN SYNDROME -axial instability, uncorrected vision or orthopedic surgery. Using lottery method, the participants will be randomly divided in to two groups. One group will be given Cuevas Medek Exercises and the other with Rebound exercises. SAMU-Disability Fitness (DISFIT) battery will be used to assess the Physical Fitness in Down syndrome. Both groups will be given three treatment session per week for 12 weeks and total time for each session will be 30-45 minutes. Data will be analyzed by using SPSS v 26.Sample size is 24 and is calculated by epitool

ELIGIBILITY:
Inclusion Criteria:

* Children with Down syndrome
* Age 3-8 years Both genders
* Children who were able to understand the commands given to them.
* They were able to stand and walk independently.

Exclusion Criteria:

* Patients with medical conditions that would severely limit their participation in the study
* Hearing loss
* Contracture
* Musculoskeletal disorders,
* Atlanto-axial instability
* Cardiac anomalies
* Thyroid abnormality
* Seizures
* Uncorrected vision problems
* Orthopedic surgery or spasticity-reduction intervention

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
SAMU-DISFITT Battery for Physical fitness | Baseline,12 weeks
  The SAMU-DISFIT battery is a reliable and feasible physical fitness battery which has been created with the purpose of establishing tests which measure the four basic components of PF (flexibility, cardiorespiratory fitness, musculoskeletal fitness and motor fitness) in DS. physical fitness (PF) of child with DS: Body Mass Index (BMI), Waist Circumference

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Afzal, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Muhammad Nouman Ashraf, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cabeza-Ruiz R, Alcantara-Cordero FJ, Ruiz-Gavilan I, Sanchez-Lopez AM. Feasibility and Reliability of a Physical Fitness Test Battery in Individuals with Down Syndrome. Int J Environ Res Public Health. 2019 Jul 27;16(15):2685. doi: 10.3390/ijerph16152685. PMID 31357594